CLINICAL TRIAL: NCT04879758
Title: The Effect of Communicating Genetic Risk of Type 2 Diabetes and Wearable Technologies On Objectively Measured Behavioral Outcomes: A Randomized Controlled Study
Brief Title: Intervention Study: Genetic Risk Communication and Wearables
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Kim, Youngwon, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: geneticriskwearabletrial
Record Dates: First submitted 2021-04-27; First posted 2021-05-10 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Fitness Trackers; Sedentary Behavior; Exercise; Genetic Predisposition to Disease; Type 2 Diabetes
Keywords: diabetes; physical activity; genetic risk; wearable technology; randomized controlled trial; movement behavior; nutrition
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Genetic Predisposition to Disease; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: parallel-group, open randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Group allocation will be concealed from study staff until the 7-day pre-intervention period begins (for preparation of corresponding e-leaflets, genetic risk estimates and/or baseline Fitbit step goal calculations), and from participants until the interventions are delivered. Given the nature of the interventions delivered, it will be impossible for participants to be blinded to the specific intervention they receive once the initial interventions are provided; however, study staff analyzing participants' de-identified data will remain blinded to participant randomization assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The control group will receive a Fitbit device and general lifestyle advice e-leaflet, which includes information about T2D, health impacts of T2D and lifestyle advice on 4 major risk markers of T2D (e.g., PA, diet, smoking, weight management) as recommended by the World Health Organization.
- Intervention Group - Genetic Risk Estimate (Experimental): This intervention group will receive an estimated genetic risk of T2D in addition to the Fitbit and e-leaflet.
  Interventions: Genetic: Genetic Risk Estimate
- Intervention Group - Genetic Risk Estimate + Fitbit Functions (Experimental): This intervention group will receive a Fitbit device, but have a Fitbit step goal set 10% higher than their baseline step count, and use its prompt functions, in addition to the genetic risk estimate and e-leaflet.
  Interventions: Other: Genetic Risk Estimate + Fitbit Functions

INTERVENTIONS:
Genetic: Genetic Risk Estimate — The genetic risk information includes individual remaining-lifetime and 10-year genetic risk estimates for T2D as well as a dichotomized genetic risk category: 'increased genetic risk' (if their genetic risk is higher than the average population risk) or 'no increased genetic risk' (if their genetic risk is not higher than the average population risk).
  Arms: Intervention Group - Genetic Risk Estimate
Other: Genetic Risk Estimate + Fitbit Functions — The genetic risk information includes individual remaining-lifetime and 10-year genetic risk estimates for T2D as well as a dichotomized genetic risk category: 'increased genetic risk' (if their genetic risk is higher than the average population risk) or 'no increased genetic risk' (if their genetic risk is not higher than the average population risk).
  The two unique Fitbit functions are step goal setting and prompts. Individualized daily step goals will be set to be 10% higher than participants' own baseline Fitbit step counts. The 'Reminder To Move' function of Fitbit will be used as a prompt to remind participants to reduce sedentary time and walk at least 250 steps/hour within a specified timeframe (i.e., from 9am to 10pm in the proposed research). If the user has not accumulated at least 250 steps/hour, a reminder (for example, 150 steps to go) will appear on the Fitbit screen at 10 minutes before the hour (for example, at 10:50 a.m.) and cause the device to vibrate.
  Arms: Intervention Group - Genetic Risk Estimate + Fitbit Functions

SUMMARY:
This study aims to determine the effects of communicating genetic risk for type 2 diabetes (T2D) alone or in combination with goal setting and prompts from a wearable device on objectively measured physical activity (PA) and sedentary behavior (SB) in East Asians. It is hypothesized that this combination will lead to significant favorable changes in objectively measured PA and SB, and that such changes will be more likely to be sustained over 6-month follow-up.

This study aims to recruit 150 healthy East Asian adults in Hong Kong. At baseline, participants will be invited to visit the research laboratory for measurement of a series of variables including height, body weight, blood pressure and grip strength. Participants will also be invited to complete a set of questionnaires to assess their self-reported PA and SB, fruit and vegetable consumption, smoking status and psychological variables. Blood samples will be collected to analyze key diabetes and cardiovascular disease biochemical markers as well as their estimated genetic risk of T2D. Each individual's unique genetic risk for T2D will be estimated on the basis of established genetic variants associated with T2D specifically for East Asians. Each participant will be asked to wear a Fitbit Charge 4 tracker, an objective activity monitoring device, throughout the entire trial.

Participants will be randomly allocated into 3 groups: 1 control and 2 intervention groups. A control group will receive an e-leaflet containing general lifestyle advice for prevention of T2D. An intervention group will receive an estimated genetic risk of T2D, in addition to the e-leaflet. The other intervention group will have a Fitbit step goal set 10% higher than their baseline step count and use prompt functions of the Fitbit tracker, in addition to the genetic risk estimate and e-leaflet.

Activity data from the Fitbit will be collected at 4-week post-intervention; information about lifestyle and psychological variables will be assessed through the questionnaires at both immediate and 4-week post-intervention. To determine the longer-term effect of the intervention, participants will be asked to visit the research laboratory 6 months after the intervention to repeat the same set of assessments as baseline, except the blood samples collected at 6-month follow-up are used only to analyze cardiometabolic risk profiles (not genetic risk). Activity levels will also be objectively measured using the Fitbit for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* East Asian ancestry
* Aged 40-60 years
* Able to perform daily-living physical activity
* Able to use English to communicate
* Use a smartphone

Exclusion Criteria:

* have been diagnosed with any type of diabetes
* pregnant or lactating
* unable to perform daily-life physical activities (determined through Physical Activity Readiness Questionnaire [PAR-Q])
* participating in another research study or exercise programs
* had experience of genetic testing
* cannot use English

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Changes in Steps between baseline and 4-week post-intervention, and between baseline and 6-month follow-up | Baseline, 4-week post-intervention, 6-month follow-up
  Step count (per day) will be objectively measured by the Fitbit tracker.
Changes in Sedentary Minutes between baseline and 4-week post-intervention, and between baseline and 6-month follow-up | Baseline, 4-week post-intervention, 6-month follow-up
  Sedentary Minutes (per day) will be objectively measured by the Fitbit tracker.
Changes in Lightly Active Minutes between baseline and 4-week post-intervention, and between baseline and 6-month follow-up | Baseline, 4-week post-intervention, 6-month follow-up
  Lightly Active Minutes (per day) will be objectively measured by the Fitbit tracker.
Changes in Fairly Active Minutes between baseline and 4-week post-intervention, and between baseline and 6-month follow-up | Baseline, 4-week post-intervention, 6-month follow-up
  Fairly Active Minutes (per day) will be objectively measured by the Fitbit tracker.
Changes in Very Active Minutes between baseline and 4-week post-intervention, and between baseline and 6-month follow-up | Baseline, 4-week post-intervention, 6-month follow-up
  Very Active Minutes (per day) will be objectively measured by the Fitbit tracker.
Changes in Calories Burn between baseline and 4-week post-intervention, and between baseline and 6-month follow-up | Baseline, 4-week post-intervention, 6-month follow-up
  Calories Burn (kcal per day) will be objectively measured by the Fitbit tracker.

SECONDARY OUTCOMES:
Changes in body mass index (BMI) between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Measured height (in meters) and body weight (in kilograms) will be used to calculate BMI (in kg/m²).
Changes in systolic blood pressure between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Systolic blood pressure (mm Hg) will be measured using the OMRON HEM-907 Digital Automatic Blood Pressure Monitor.
Changes in diastolic blood pressure between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Diastolic blood pressure (mm Hg) will be measured using the OMRON HEM-907 Digital Automatic Blood Pressure Monitor.
Changes in hand grip strength between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Hand grip strength (in kilograms) will be measured using the Jamar Hydraulic Hand Dynamometer, which has good reliability and reproducibility.
Changes in Hemoglobin A1c (HbA1c) between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Blood samples will be collected to test the five key biochemical markers of T2D and cardiovascular disease, including HbA1c (%).
Changes in Total cholesterol between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Blood samples will be collected to test the five key biochemical markers of T2D and cardiovascular disease, including Total cholesterol (mmol/L).
Changes in High-density lipoproteins (HDL) between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Blood samples will be collected to test the five key biochemical markers of T2D and cardiovascular disease, including HDL (mmol/L).
Changes in Low-density lipoproteins (LDL) between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Blood samples will be collected to test the five key biochemical markers of T2D and cardiovascular disease, including LDL (mmol/L).
Changes in Triglycerides between baseline and 6-month follow-up | Baseline and 6-month follow-up
  Blood samples will be collected to test the five key biochemical markers of T2D and cardiovascular disease, including Triglycerides (mmol/L).
Changes in Self-reported Physical Activity between baseline and Immediate post-intervention, between baseline and 4-week post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 4-week post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.
Changes in Self-reported Fruit and Vegetable Consumption between baseline and Immediate post-intervention, between baseline and 4-week post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 4-week post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.
Changes in Self-reported Smoking Status between baseline and Immediate post-intervention, between baseline and 4-week post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 4-week post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.
Changes in Self-reported Psychological Status between baseline and Immediate post-intervention, between baseline and 4-week post-intervention, and between baseline and 6-month follow-up | Baseline, Immediate post-intervention, 4-week post-intervention, 6-month follow-up
  This outcome will be assessed using an assessment questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Youngwon Kim, Principal Investigator — The University of Hong Kong
Locations (1):
- Exercise Physiology Lab, The University of Hong Kong, Hong Kong, Hong Kong